CLINICAL TRIAL: NCT00846560
Title: Involvement of Lymphocyte Type B in Amyotrophic Lateral Sclerosis (ALS)
Status: Withdrawn | Type: Observational
Why Stopped: Changes in the lab's focus and needs
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, d_yarnitsky, Head of Neurology Department, Rambam Health Care Campus
Other Study IDs: ALS04CTIL
Record Dates: First submitted 2009-02-15; First posted 2009-02-18 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 ALS patients
- 2 Healthy subjects

SUMMARY:
The involvement of Lymphocyte type B in Amyotrophic lateral sclerosis (ALS) patients will be compared to lymphocyte in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients who could sign ICF.

Exclusion Criteria:

* No ALS patients age less than 18 years.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Amyotrophic lateral sclerosis and Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical center, Neurology Department, Haifa, Israel